CLINICAL TRIAL: NCT06551922
Title: Effects of Instrumental Soft Tissue Mobilization Technique With and Without Conservative Treatment on Pain , Range of Motion and Functional Disability in Post Operative Knee Stiffness Patients
Brief Title: Effects of IASTM With and Without CT on Pain, ROM, and Functional Disability in Post-Operative Knee Stiffness Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Sawera Ali, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-/198/08/24
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Pain; Pain, Postoperative; Pain, Joint; Knee Pain Chronic
Keywords: Range of motion; Knee Stiffness; Functional Disability; Conservative treatment; Instrument-Assisted Soft Tissue Mobilization
MeSH Terms: conditions — Pain; Pain, Postoperative; Arthralgia | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: * Group A (Instrumental Soft Tissue Mobilization Technique with Conservative Treatment)
  * Group B (Conservative Treatment Only)
Who Masked: Outcomes Assessor
Masking Description: The single-blinded assessor was utilized to minimize bias in outcome measurements. The assessor was unaware of the intervention group assignment for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrumental Soft Tissue Mobilization Technique with Conservative Treatment (Experimental): Apply TENS for 10 minutes to administer a microcurrent therapy to participants. The IASTM was applied for 90 seconds- 2 minutes on each muscle along with the stretching exercises. The intervention was applied 3 times per week.
  Muscle involved:
  * Hip Adductors
  * Hamstrings
  * Quadriceps
  * Patellar tendon
  * Iliotibial band
  * Calf muscles.
  Interventions: Combination Product: Instrumental Soft Tissue Mobilization Technique with Conservative Treatment
- Conservative Treatment (Experimental): For conservative treatment apply TENS for 10 minutes to administer a micro current therapy to participants. Than Stretching exercises ( Hamstrings and Quadriceps), Strengthening exercises (Quadriceps, Hamstring, Calf ), Balance exercises and Ice Therapy.
  Interventions: Combination Product: Conservative Treatment

INTERVENTIONS:
Combination Product: Instrumental Soft Tissue Mobilization Technique with Conservative Treatment — TENS: Apply TENS for 10 minutes on the greater trochanter and the area just above the lateral knee joint line, adhesive electrodes were positioned.
  Frequency: 3 times per week. Duration: 90 seconds- 2 minutes on each muscle (Purbia, 2023). Technique: A therapist uses Ergon tools to apply gentle pressure and strokes along the targeted muscles and fascial tissues. Different IASTM techniques, like stroking, raking, and hooking, address specific tissue restrictions. The therapist should continue the IASTM technique for 5-10 minutes, or until the stiffness in the knee is reduced (Mubashar et al., 2022; Purbia, 2023).
  Conservative Treatment: Stretching exercises for the hamstrings and quadriceps to improve flexibility and reduce tension. Affected iliotibialband. Hold for 30 seconds. Uncross your legs and stand up straight again. Repeat four more times (Mubashar et al., 2022).
  Arms: Instrumental Soft Tissue Mobilization Technique with Conservative Treatment
Combination Product: Conservative Treatment — TENS: Apply TENS for 10 minutes on the greater trochanter and the area just above the lateral knee joint line, adhesive electrodes were positioned.
  Stretching exercises with hold for 30 seconds. Uncross your legs and stand up straight again (Mubashar et al., 2022).
  Quadriceps Strengthening: Perform exercises like straight leg raises, seated leg press and squats to strengthen (Lim & Al-Dadah, 2022).
  Hamstring Strengthening: Include exercises like leg curls to strengthen the hamstring muscles (Lim & Al-Dadah, 2022).
  Calf Strengthening: Perform calf raises to strengthen the calf muscles (Lim & Al-Dadah, 2022).
  Balance Exercises: Incorporate balance exercises like single-leg stands on a foam pad (Lim & Al-Dadah, 2022).
  Ice Therapy: Apply ice packs to the affected knee for 15-20 minutes (Lim & Al-Dadah, 2022).
  Arms: Conservative Treatment

SUMMARY:
This single-blinded randomized control study aimed to determine the effects of instrumental soft tissue mobilization technique with and without conservative treatment in post-operative knee stiffness patients. This study recruited 84 participants who fulfilled the inclusion criteria and were randomly divided into experimental and control groups using the lottery method. The assessor was unaware of the treatment given to both groups. Data were collected at baseline, at the end of the third week, and at the end of the sixth week. Baseline assessments were conducted before the intervention. Post-intervention assessments were conducted immediately after the intervention. This study aimed to investigate the effectiveness of IASTM, both with and without traditional conservative treatment methods, in improving pain, range of motion, and functional ability in patients experiencing post-operative knee stiffness. By examining these factors, we gained valuable insights into the potential of IASTM as a therapeutic intervention for this challenging condition.

DETAILED DESCRIPTION:
Instrument-Assisted Soft Tissue Mobilization (IASTM) is emerging as a valuable tool for physiotherapists, offering a range of benefits for both practitioners and patients. By integrating IASTM with traditional methods, physiotherapists can elevate the standard of care, improve patient outcomes, and even contribute to a healthier community.

Study Design:

* Randomized Control Trial

Screening:

* Patients were screened to meet inclusion criteria. The consent form was taken from patients and then randomly allocated into two groups ( 42 in each group).

Randomization:

* Patients fulfilling the inclusion criteria were randomly divided into experimental and control groups using the lottery method.

Blinding:

* The study was single-blinded. The assessor was unaware of the treatment given to both groups.

Assessment:

* Data was collected at baseline, at the end of the third week and the end of 6th week. Baseline assessments were conducted before the intervention. Post-intervention assessments were conducted immediately after the intervention.

Intervention:

* Group A (Instrumental Soft Tissue Mobilization Technique with Conservative Treatment)
* Group B (Conservative Treatment Only)

Progress Monitoring:

* Treatment intensity and exercise difficulty were progressively adjusted for both groups throughout the intervention based on participant tolerance and progress.

Ethical Considerations:

* This study has received ethical approval from the Institutional Review Board (IRB). Informed consent was obtained from all participants.

Data Analysis:

* Statistical software was used to analyze the data, with appropriate tests employed based on data normality to compare outcomes between groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 25 to 50 years (Meena et al., 2023)
* Participants of both genders (Meena et al., 2023)
* Participants who have undergone post-operative knee stiffness surgery (Meena et al., 2023)
* Patients having knee fracture (Poliakov et al., 2020).

Exclusion Criteria:

* Patients with total knee replacement (Poliakov et al., 2020).
* Participants with knee osteoarthritis or other knee conditions not related to post-operative knee stiffness (Meena et al., 2023)
* Participants with other joint conditions not related to the knee (Mezey et al., 2023)
* Post-operative knee stiffness patients with comorbidities that may affect the outcome of the study (Mezey et al., 2023)

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2024-01-28 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 6 weeks (baseline, third week and then at the end of the sixth week)
  Pain level measured using a visual analog scale. It consists of a 10-centimeter line with endpoints labeled to represent the two extremes of the experience being measured. For pain, the typical endpoints are "no pain" on the left and "worst imaginable pain" on the right. For pain, a score of 0 means no pain, while a score of 10 represents the worst imaginable pain.
Range of motion | 6 weeks (baseline, third week and then at the end of the sixth week)
  Range of motion measured using a goniometer

SECONDARY OUTCOMES:
Functional disability | 6 weeks (baseline, third week and then at the end of the sixth week)
  Functional disability measured using the Lower Extremity Functional Scale. The scale consists of 20 items that assess the patient's ability to perform various activities, such as walking, running, and climbing stairs. The objective of the LEFS is to measure patients' initial function, ongoing progress, and outcome for a wide range of lower-extremity conditions. The maximum total score is 80, indicating no functional limitations.The minimum score is 0, indicating extreme limitations. The lower the total score, the greater the disability

CONTACTS AND LOCATIONS:
Overall Officials: Asim Arif, M.Phil MSK, Principal Investigator — University of Lahore; Alishba Mustansar, M.Phil./tDPT, Study Director — University of Lahore
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mubashar, H., Hassan, D., & Bushra, M. (2022). Effects of Instrumented Assisted Soft Tissue Mobilization (IASTM) Technique Versus Stretching on Ililotibal Band in Patients with Anterior Knee Pain. Pakistan Journal of Medical & Health Sciences, 16(11), 353-353.
- [Background] Poliakov, A., Pakhaliuk, V., & Popov, V. L. (2020). Current trends in improving of artificial joints design and technologies for their arthroplasty. Frontiers in Mechanical Engineering, 6, 4.
- [Background] Purbia, C. (2023). Effectiveness of KIASTM technique applied only quadriceps muscle for knee pain. International Journal of Orthopaedics, 9(3), 379-383.
- [Result] Lim WB, Al-Dadah O. Conservative treatment of knee osteoarthritis: A review of the literature. World J Orthop. 2022 Mar 18;13(3):212-229. doi: 10.5312/wjo.v13.i3.212. eCollection 2022 Mar 18. PMID 35317254
- [Result] Meena A, Hoser C, Abermann E, Hepperger C, Raj A, Fink C. Total knee arthroplasty improves sports activity and the patient-reported functional outcome at mid-term follow-up. Knee Surg Sports Traumatol Arthrosc. 2023 Mar;31(3):905-913. doi: 10.1007/s00167-022-07025-z. Epub 2022 Jun 11. PMID 35689683
- [Result] Cutie MR, Lordi NG. Compatibility of verapamil hydrochloride injection in commonly used large-volume parenterals. Am J Hosp Pharm. 1980 May;37(5):675-6. PMID 7386476